CLINICAL TRIAL: NCT00431873
Title: A Phase II Study of MGCD0103 (MG-0103) in Patients With Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-009
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Lymphocytic Leukemia, Chronic
Keywords: Lymphocytic Leukemia, Chronic (Refractory); Phase II
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Lymphoid; Bronchiolitis Obliterans Syndrome | interventions — mocetinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MGCD0103 administered orally three times per week.
  Interventions: Drug: MGCD0103

INTERVENTIONS:
Drug: MGCD0103 — MGCD0103 Administered orally three times per week.

SUMMARY:
In this study, MGCD0103, a new anticancer drug under investigation, is given three times weekly to patients with refractory chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of CLL.
* Prior Treatment. There will be no limit to prior therapy. Therapy with fludarabine and Rituxan must have failed (disease progression, intolerance, or not a candidate).
* Age 18 years or greater.
* ECOG performance status of 0 or 1.
* Laboratory requirements (must be done within 7 days prior to study initiation):

  * Total Bilirubin ≤ 1.5 x Upper Limit of Normal (ULN).
  * Aspartate transaminase (AST/SGOT) and Alanine transaminase (ALT/SGPT) ≤ 2.5 x ULN.
  * Serum Creatinine ≤1 .5 x ULN.
* Patients or their legal representative must be able to read, understand, and sign a written informed consent (approved by the institutional review board/Ethics Committee (IRB/EC)) within 14 days prior to start of treatment.

Exclusion Criteria:

* Patients with another active cancer (excluding basal cell carcinoma or cervical intraepithelial neoplasia (CIN/cervical in situ) or melanoma in situ). Prior history of cancer is allowed, as long as there is no active disease.
* Pregnant or lactating women. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test documented within 7 days prior start of study drug.
* WOCBP and men whose partners are WOCBP must use an acceptable method of contraception while enrolled on this study, and for a period of 3 months following study drug treatment. Patients unwilling or unable to follow this guideline will be excluded. An example of an acceptable form of contraception is a double barrier method, such as condom with diaphragm.
* Patients with uncontrolled intercurrent illness, active or uncontrolled infections, or a fever > 38.5ºC (not due to tumor fever) on the day of scheduled dosing.
* Patients with serious illnesses, medical conditions, or other medical history, including laboratory results, which, in the investigator's opinion, would be likely to interfere with a patient's participation in the study, or with the interpretation of the results.
* Patients who have been treated with any investigational drug within 28 days prior to study initiation (an investigational drug is one for which there is no approved indication), or who are receiving concurrent treatment with other experimental drugs or anti-cancer therapy. Patients must have recovered from all transient toxicity induced by prior therapy.
* Known hypersensitivity to HDAC inhibitors, to any of the components of MG-0103 (refer to IB). Patients who have known anaphylaxis or IgE-mediated hypersensitivity to murine proteins or to any component of rituximab will not be allowed to receive rituximab concomitantly on this study.
* Known human immunodeficiency virus (HIV) or known active Hepatitis B or C. Testing is not required for patients not suspected of having these conditions. For patients with a history of Hepatitis B or C that is no longer active, the Investigator should contact MethylGene in advance to confirm patient's eligibility.
* Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location, etc) that, in the judgment of the investigator, may affect the patient's ability to sign the informed consent and undergo study procedures.
* Any condition that will put the patient at undue risk or discomfort as a result of adherence to study procedures. For example, consider requirement to take MG-0103 with a low-pH drink and recommendation to avoid agents that increase gastric-pH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Response rate | 1 year (anticipated)

SECONDARY OUTCOMES:
Duration of objective response | 1 year (anticipated)
Safety profile | 1 year (anticipated)
Pharmacodynamics (biomarkers) | 1 year (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (13):
- United States (6):
  - Veteran Affairs Medical Center Research Service, Kansas City, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic/Chronic Leukemia/Multiple Myeloma Program, Cleveland, Ohio
  - Ohio State University, James Cancer Hospital, Colombus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Canada (7):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster University Health Center, Hamilton, Ontario
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - UHN - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles-LeMoyne, Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHA, Hopital Enfant-Jesus, Québec, Quebec